CLINICAL TRIAL: NCT01162629
Title: An Evaluation of Vertical Augmentation of Alveolar Bone With Osteon at Dental Implant Placement
Brief Title: Vertical Augmentation With Osteon at Dental Implant Placement
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Research and Education in Dentistry (Other)
Responsible Party: Dr Richard Oliver, Research and Education in Dentistry
Other Study IDs: RED001
Record Dates: First submitted 2010-07-05; First posted 2010-07-14 (Estimated); Last update posted 2010-07-15 (Estimated); Status verified 2010-07

CONDITIONS: Tooth Injuries; Tooth Abnormalities
Keywords: bounded saddles; missing teeth; dental implants; Tooth, Nonvital
MeSH Terms: conditions — Tooth Injuries; Tooth Abnormalities; Anodontia; Tooth, Nonvital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Osteon: Patients requiring dental implants with deficient alveolar bone height
  Interventions: Device: Osteon bone graft

INTERVENTIONS:
Device: Osteon bone graft — Osteon bone substitute placed to a height of 2 mm above the top of the dental implant
  Other Names: Osteon; Hydroxyapatite coated with beta-tricalcium phosphate; 100% synthetic bone graft

SUMMARY:
Dental implants are a valid and reliable method to replace missing teeth. The major requirement for their success is an adequate volume of bone into which they can be placed. One widely used method to augment bone at the time of placing the implant is to use a bone substitute rather than taking a block bone graft from the patient. Successful augmentation in the vertical direction has often proved difficult, however, the investigators have developed a technique to achieve this in the investigators patients using a synthetic bone substitute, Osteon (Implantium, CE0120) in an attempt to avoid patients having to undergo another unnecessary surgical procedure.

DETAILED DESCRIPTION:
Primary Objective

• To determine the success of dental implants in alveolar bone augmented in the vertical direction with Osteon.

Secondary Objectives • To determine the long term success of dental implants in this augmented bone.

Primary Endpoint

• Radiographically assessed vertical height of alveolar ridge formation following Osteon augmentation.

ELIGIBILITY:
Inclusion Criteria:

* missing one or two teeth
* bounded saddle
* healthy (ASA grade I & II) adult

Exclusion Criteria:

* smoker
* significant medical problem (ASA III or above)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Private specialist dental implant clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
The success of dental implants in alveolar bone augmented in the vertical direction with Osteon | 3 years
  The implants will be deemed successful at each time point if the radiographic bone level remains at 2 mm above the level of the implant, i.e. at the same height as when placed. Given that we know precisely the dimensions of the abutments placed in the implant, this provides the necessary calibration in order to undertake this assessment. If the bone level is lost, the procedure will be deemed to have failed.

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Oliver, BDS PhD, Principal Investigator — Research and Education in Dentistry
Locations (1):
- Oracle Dental Clinics, Shrewsbury, Shropshire, United Kingdom